CLINICAL TRIAL: NCT05587582
Title: Behavioral Parenting Skills as a Novel Target for Improving Pediatric Medication Adherence: Studies 1 and 2
Brief Title: Behavioral Parenting Skills As A Novel Target for Improving Pediatric Medication Adherence
Status: Completed | Type: Observational
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: I 1832021; R01CA258337 (NIH)
Record Dates: First submitted 2022-10-14; First posted 2022-10-20 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (Family Behaviors): PRIMARY OBJECTIVES:
  I. Use direct observation of medication administration in the home to understand common episode-level barriers and identify the most impactful behavioral parenting skills for intervention.
  II. Use daily diary methods to identify contextual barriers to adherence and identify intervention components to help parents anticipate barriers and plan strategies to promote successful adherence.
  OUTLINE:
  Participants complete a survey over 15-20 minutes at baseline. Family behaviors before, during and after the administration of medication to the child are video-recorded over 40-45 minutes. Participants receive MEMS electronic pill bottle to use for 2 weeks and complete daily survey over 5 minutes for 14 days.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete a survey

SUMMARY:
This study observes behavioral parenting skills to see whether it could be a novel target for improving pediatric medication adherence. This study may help researchers better understand the challenges parents face when giving their young child with an illness medicine at home and learn about various factors related to medication compliance in young children

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Use direct observation of medication administration in the home to understand common episode-level barriers and identify the most impactful behavioral parenting skills for intervention.

II. Use daily diary methods to identify contextual barriers to adherence and identify intervention components to help parents anticipate barriers and plan strategies to promote successful adherence.

OUTLINE:

Participants complete a survey over 15-20 minutes at baseline. Family behaviors before, during and after the administration of medication to the child are video-recorded over 40-45 minutes. Participants receive MEMS electronic pill bottle to use for 2 weeks and complete daily survey over 5 minutes for 14 days.

ELIGIBILITY:
INCLUSION:

* Parent of a child diagnosed within the past month with acute lymphoblastic leukemia (ALL)
* Pediatric patient's age 3 - 9.

  * If present during the home visit, any other child, ages 0-18
* Child on therapy that includes oral mercaptopurine (6-MP) administration
* Parent age 18 - NA (No Limit)
* Parent should have verbal English fluency
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* The following special populations may be included in this study:

  * Pregnant women: due to the design of this behavioral research, pregnant and fetuses should incur no elevated risk from participation.

Children under age 18 will participate in one aspect of the study, the video recording of medication administration.

* Other children (not the pediatric patient) under age 18 that are present during the time of the home visit

Exclusion:

* Pediatric patient is on therapy that does not include oral 6-MP administration
* Cognitively impaired adults/adults with impaired decision-making capacity
* Pediatric patients who are not yet adults (infants under the age of 3, children over 9 years, teenagers)
* Prisoners

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Families of young children ages 3-9 diagnosed with acute lymphoblastic leukemia within 4 weeks of oral chemotherapy prescription at Roswell Park Cancer Institute (Buffalo, NY) or Oishei Children's Hospital in Buffalo, New York
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Dyadic Parent-Child Interaction Coding System (DCIPS) - medication ingestion | Up to 5 months
  Association between ingestion of medication and the absence or presence of each of the Observations of parents and children as they interact with each other during medication administration. Interactions will be coded by trained observers.
Length of time it takes to administer medication | Up to 5 months
  The association between time to ingestion and the DCIPS coded skills will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Bouchard, PhD, Principal Investigator — Roswell Park Comprehensive Cancer Center
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided